CLINICAL TRIAL: NCT00527540
Title: Effectiveness and Side Effects of Pegylated Interferon Alpha-2a (Pegaferon®) Plus Ribavirin in the Patients With Chronic Hepatitis C
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tehran Hepatitis Center (Other)
Collaborators: Kermanshah University of Medical Sciences (Other)
Responsible Party: Prof SM Alavian, Tehran Hepatitis Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: THC-10
Record Dates: First submitted 2007-09-08; First posted 2007-09-11 (Estimated); Last update posted 2009-01-21 (Estimated); Status verified 2009-01

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Pegylated Interferon alpha 2a + Ribavirin — Pegaferon: Ampule, 180 microgram per week Ribaverin: Tablet, 10-15 mg/kg per day
  Other Names: Pegaferon

SUMMARY:
Pegylation of interferon prolongs the medication half-life which has resulted in Pegylated Interferon (PEG-IFN) as the new modality for treatment of chronic hepatitis C. We current this clinical trial to assess the efficacy and safety of domestic PEG-IFN alpha-2a (Pegaferon®) in the patients with chronic hepatitis C.

DETAILED DESCRIPTION:
We enroll 50 patients in to the study. The patients receive Pegaferon® 180 micgr per week plus ribavirin 10-15mg/kg per day. The patients are visited every 4 weeks with biochemistry lab tests. They are checked with quantitative HCV PCR on the third month after initiation of the treatment to assess early virologic response and at the end of the study for complete response rate and on the six month after treatment completion for sustained response rate. The patients with undetectable HCV RNA are considered as responders.

ELIGIBILITY:
Inclusion Criteria:

* HCV RNA: Positive
* Biopsy approved in genotype 1
* Age older than 18 yrs

Exclusion Criteria:

* ongoing pregnancy or breast feeding
* Hx of hemochromatosis
* Hx of metabolic liver dis.
* Hx of HCC
* Hx of autoimmune hepatitis
* Hx of alcoholic liver dis.
* Hx of bleeding from esophageal varices
* ongoing systemic anti-viral or anti-neoplasmic treatment
* Hx of treatment with an anti-depressant medication at therapeutic doses for at least 3 months at any pervious time
* Hx of treatment with an tranquilizer at therapeutic doses for psychosis for at least 3 months at any pervious time
* Hx of hospitalization for psychiatric dis.
* Hx of suicidal attempt
* Hx of IBD
* Hx of SLE
* Hx of scleroderma
* Hx of rheumatoid arthritis
* Hx of ITP
* Hx of autoimmune hemolytic anemia
* Hx of severe psoriasis
* Hx of chronic pulmonary dis. associated with functional limitation
* Hx of MI or unstable angina
* Hx of arrhythmia requiring ongoing treatment
* Hx of functional class III or IV
* Hx of severe seizure dis. or current anti-convulsant use
* Hx of organ transplantation with existing functional graft
* Hx of severe retinopathy
* Hx of Thalassemia
* Hx of spherocytosis
* Hx of cerebrovascular dis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2007-02; Primary Completion 2008-06 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
End of treatment response rate (HCV RNA:Neg) | End of treatment course

SECONDARY OUTCOMES:
Sustain response rate (HCV RNA:Neg) 6 month after end of treatment | 6 month after end of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Seyed M Alavian, Prof., Study Chair — Tehran Hepatitis Center; Behzad Hajarizadeh, MD, Principal Investigator — Tehran Hepatitis Center
Locations (1):
- Tehran Hepatitis Center, Tehran, Tehran Province, Iran